CLINICAL TRIAL: NCT06333938
Title: An Effectiveness-Implementation Hybrid Study on the Use of Integrative Treatments for Perioperative Symptom Management.
Brief Title: Veterans Enhanced Recovery Using Integrative Treatments Around Surgery
Acronym: VERITAS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01968
Record Dates: First submitted 2023-12-13; First posted 2024-03-27 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Surgery; Knee Arthropathy
Keywords: Perioperative Care; Complementary Integrative Health (CIH); Battlefield Acupuncture (BFA); Music Medicine; Aromatherapy; Veterans; Integrative Treatments
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrative Treatment (Active Comparator): 200 participants will receive at least one of three integrative treatments: Music Medicine, Aromatherapy, Battlefield Acupuncture
  Interventions: Other: Nonpharmacologic Treatment
- Standard Care (Active Comparator): 200 patients will not receive standard care without any additional integrative treatments
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Nonpharmacologic Treatment — At least one three nonpharmacologic treatments (Music Medicine, Aromatherapy, Battlefield Acupuncture) will be delivered. Music Medicine is the delivery of personal music players to listen to patient-preferred music before, during, or after surgical or non-surgical procedures. Aromatherapy is the delivery of personally-preferred AromaTabs before, during, or after surgical or non-surgical procedures. Battlefield Acupuncture is the delivery of Auricular Acutherapy by trained providers using acupuncture needles or acupressure beads before, during, or after surgical or non-surgical procedures.
  Arms: Integrative Treatment
Other: Standard Care — Patients will receive standard clinical care without the addition of Music Medicine, Aromatherapy, or Battlefield Acupuncture
  Arms: Standard Care

SUMMARY:
The study aims to assess the implementation and effectiveness of Integrative Treatments - Music Medicine, Aromatherapy, and Battlefield Acupuncture - in the management of perioperative pain and anxiety, and in the reduction of related pharmacologic treatments.

DETAILED DESCRIPTION:
There is an urgent need for effective, safe, and low-cost nonpharmacologic treatments for postoperative pain. This study aims to:

1. assess the implementation of Music Medicine, Aromatherapy, and Battlefield Acupuncture among patients presenting for procedures at the Durham Veterans Affairs Medical Center; and,
2. compare the effectiveness of these treatments, alone and in combination, versus standard clinical practice not involving any of these treatments.

Patients from the Durham Veterans Affairs Medical Center (Durham VAMC) scheduled to undergo procedures will be eligible to participate in this study. A sample of 400 veterans will be studied. We will offer treatments versus no treatment on alternate months. Recruitment will end when 200 patients have received at least one of these treatments, and 200 patients have received no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans Scheduled to undergo procedures at the Durham VA

Exclusion Criteria:

* Hearing Loss
* Procedures on the Ear
* Risk of Bleeding
* Anosmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Pain and Pain Interference assessed among patients using the Defense veterans pain rating scale 2.0 | Each day from Postoperative Day 0 to Day 5.
  The Defense and Veterans Pain Rating Scale 2.0 utilizes a numerical rating scale enhanced by functional word descriptors, color coding, and pictorial facial expressions matched to pain levels. Four supplemental questions measure how much pain: a) interferes with usual activity, b) interferes with sleep, c) affects mood and d) contributes to stress. The scale for each assessment ranges from 0-10. Three assessments will occur each day. The daily average values will be compared at each time point. Higher Scores represent worse outcomes.
Heart Rate Variability among Patients as assessed using time and frequency domain analysis of the heart rate. | Each day (over 8-hour periods, 7pm and 7am) from 5 days before surgery to postoperative day 5.
  Heart rate variability represents the change in the time interval in milliseconds between successive heartbeats. It is a measure of input to the heart from both sympathetic and parasympathetic branches of the nervous system. Increased heart rate variability is the better outcome.
Implementation of Treatment among Patients as assessed by the Acceptability of Intervention, Appropriateness of Intervention, and Feasibility of Intervention Measures. | Measurement will be at three points: within the 5 day period before surgery; on the day of Surgery; and on postoperative day 5.
  The Acceptability of Intervention measure, Appropriateness of Intervention measure, and Feasibility of Intervention Measure will be used. Each of these three tools is a 4-item questionnaire that has been validated as a distinct and strong measure of implementation success. Scale values for each measure range from 1-5. The average of the three measures will be computed and compared at each time point. Higher scores represent better outcomes.
Fidelity of Treatment among Patients as assessed by a Fidelity Checklist | Each day from Postoperative Day 0 to Day 5.
  Fidelity, the degree to which an intervention was implemented as it was intended by the developers, will be measured using a fidelity instrument with three domains: adherence (adherence to each component of treatment, scale 1- 5), participant responsiveness (measured on the treatment expectation questionnaire scale 0-10), and dosage (scale 1-5). Higher scores are better. We will compare the average scores overall, and in each domain.
Implementation of Treatment among Providers as assessed by the Acceptability of Intervention, Appropriateness of Intervention, and Feasibility of Intervention Measures. | On the day of surgery or within 1-day after.
  The Acceptability of Intervention measure, Appropriateness of Intervention measure, and Feasibility of Intervention Measure will be used. Each of these three tools is a 4-item questionnaire that has been validated as a distinct and strong measure of implementation success. Scale values for each measure range from 1-5. The average of the three measures will be computed and compared. Higher scores represent better outcomes.
Fidelity of Treatment among Providers as assessed by a Fidelity Checklist | On the day of surgery or within 1-day after.
  Fidelity, the degree to which an intervention was implemented as it was intended by the developers, will be measured using a fidelity instrument with two domains: adherence (adherence to each component of treatment, scale 1- 5), and participant responsiveness (measured on the treatment expectation questionnaire scale 0-10). Higher scores are better. We will compare the average scores overall, and in each domain.

SECONDARY OUTCOMES:
Amount of Opioid medication received by patients assessed in average daily oral morphine equivalents. | Each day from Postoperative Day 0 to Day 5.
  The amount of opioid analgesic medications received by patients as recorded in the electronic health record (inpatient setting) or as reported by patients (outpatient setting) will be summarized each day and reported in daily oral morphine equivalents. The total amount from postoperative day 0 to day 5, and the average daily oral morphine equivalents will be measured for comparisons. Higher amounts represent worse outcomes.
Quality of Recovery among patients as measured using the Quality-of-Recovery 40 tool. | Preoperative on the day of surgery, and each day from Postoperative Day 0 to Day 5.
  The Quality-of-Recovery 40 tool is a 40-item questionnaire, with each question graded on a five-point Likert scale. Scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery). Assessment will occur preoperatively on the day of surgery (baseline value) and each day from Postoperative Day 0 to 5. The difference between the baseline and the value each day will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Durham Veterans Affairs Medical Center, Durham, North Carolina, United States